CLINICAL TRIAL: NCT03922386
Title: ProspEctive Record of Safety and Electrical Performances Of XFINE Leads: an International Study
Brief Title: Safety and Electrical Performances of XFINE Leads
Acronym: PERSEPOLIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MicroPort CRM (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LBFX05 - PERSEPOLIS
Record Dates: First submitted 2019-04-15; First posted 2019-04-22 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Intervention Model Description: Post market, multicenter, international, prospective, open label, two arms and longitudinal non comparative non randomized study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JX model (Other): Subjects implanted with an RA XFINE lead (JX model)
  Interventions: Device: XFINE leads
- TX model (Other): Subjects implanted with an RV XFINE lead (TX model)
  Interventions: Device: XFINE leads

INTERVENTIONS:
Device: XFINE leads — Pacemaker subjects with at least one XFINE passive lead

SUMMARY:
The purpose of the study is to confirm the safety and the electrical performances of the XFINE passive pacing leads, for both right ventricular (RV) straight models and right atrial (RA) J-shape models, up to 12 months follow-up post implant.

DETAILED DESCRIPTION:
All subjects will be followed until 12 months follow-up post implant.

At each follow-up visits (3, 6 and 12 months), electrical performances will be measured and safety will be monitored during the whole study duration.

ELIGIBILITY:
Inclusion Criteria:

1. Any subject newly implanted according to the most recent guidelines from the European Society of Cardiology (ESC) for less than10 days with:

   * a Single Chamber (SR) or a Dual Chamber (DR) pacemaker from Microport CRM S.r.l.
   * any right atrial and/or right ventricular XFINE lead
2. Have reviewed, signed and dated the informed consent

Exclusion Criteria:

1. Included in another clinical study that could confound the results of this study such as studies involving intra-cardiac device
2. Contraindication to a maximum single dose of 310 µg Dexamethasone Sodium Phosphate (DSP)
3. Tricuspid valvular disease or tricuspid replacement heart valve (mechanical or tissue) only for subject with DR pacemaker
4. Active myocarditis, pocket and/or lead infection
5. Age less than 18 years old or under guardianship or kept in detention
6. Life expectancy less than 1 year
7. Known pregnancy, women breastfeeding or in childbearing age without an adequate contraceptive method
8. Be unavailable for the scheduled follow-up associated with this clinical study or refusal to cooperate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-07-23 (Actual)

PRIMARY OUTCOMES:
Freedom from XFINE lead-related complications | at 6 months post implant
  This endpoint will confirm the freedom from XFINE Lead-Related Complications (LRC) up to the 6 months post implant follow-up. The anticipated complication-free rate is 0.95, and will be compared against an a priori performance goal of 0.85.
  An XFINE Lead-Related Complication (LRC) is defined as any XFINE (RA and/or RV) lead-related Serious Adverse Device Effect (SADE) that resulted in subject death or required an additional invasive intervention (excluding re-programming) and occurred within 6 months post implant. This endpoint will be assessed independently for each lead model.
Electrical performances confirmation | at 6 months post implant
  This endpoint will characterize the XFINE lead performances in ensuring adequate Pacing Capture Thresholds (PCT) through 6 months post implant follow-up. The values assessed in this analysis are the PCT measured at 0.50 ms (or less) pulse width at 6 months follow-up visit. The PCT measured at 6 months will be compared against an a priori performance goal of 1.0V/0.5 ms, assuming an expected pacing threshold at 6 months of 0.8V/0.5 ms with a standard deviation of 0.5V. This endpoint will be assessed independently for each lead model.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Bardají, Dr., Principal Investigator — Hospital Universitari Joan XXIII, Tarragona, Spain
Locations (19):
- France (3):
  - Centre Hospitalier de Cahors, Cahors
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hôpital de la Croix-Rousse, Lyon
- Italy (7):
  - Clinica Medica - Azienda Ospedaliero Universitaria Careggi, Florence
  - Ospedale Santa Maria Nuova, Florence
  - Clinica San Carlo, Milan
  - Azienda Ospedaliera Santa Maria degli Angeli, Pordenone
  - Ospedale Policlinico Casilino, Roma
  - Ospedale Civile di Vigevano, Vigevano
  - Ospedale Civile di Voghera, Voghera
- Portugal (4):
  - Centro Hospitalar do Baixo Vouga, E.P.E., Aveiro
  - Centro Hospitalar do Alto Ave - Hospital da Senhora da Oliveira, Creixomil
  - Centro Hospitalar de Leiria - Hospital de Santo André, Leiria
  - Centro Hospitalar Vila Nova de Gaia/Espinho, Vila Nova de Gaia
- Spain (2):
  - Hospital Universitari Joan XXIII, Tarragona
  - Hospital Doctor Peset, Valencia
- United Kingdom (3):
  - Leeds Teaching Hospitals NHS Trust - Leeds General Infirmary, Leeds
  - Kingston Hospital, London
  - Lister Hospital, Stevenage